CLINICAL TRIAL: NCT06090565
Title: Cefixime 800 mg Plus Doxycycline 100 mg b.i.d. for 7 Days Compared to Ceftriaxone 1 g Plus Azithromycin 2 g for Treatment of Urogenital, Rectal and Pharyngeal Gonorrhoea: A Randomised Controlled Trial
Brief Title: Cefixime Plus Doxycycline Compared to Ceftriaxone Plus Azithromycin for Treatment of Gonorrhoea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bulovka Hospital (Other)
Collaborators: Örebro University, Sweden (Other)
Responsible Party: Principal Investigator, Filip Rob MD, PhD, Head of Dermatovenereology Dept., Bulovka Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9937
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Gonorrhea
Keywords: Neisseria gonorrhoeae; Cefixime; Azithromycin; Ceftriaxone; Doxycycline
MeSH Terms: conditions — Gonorrhea | interventions — Cefixime; Doxycycline; Ceftriaxone; Azithromycin

STUDY DESIGN:
Intervention Model Description: Patients were randomised to cefixime 800 mg single oral dose plus doxycycline 100 mg twice a day orally for 7 days or the comparator ceftriaxone 1 g single intramuscular dose plus azithromycin 2 g single oral dose with a computer-generated pseudo-random code using permuted block randomisation in a 1:1 ratio
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cefixime plus doxycycline (Experimental): Single-dose cefixime 800 mg plus doxycycline 100 mg b.i.d. for 7 days
  Interventions: Drug: Cefixime; Drug: Doxycyclin
- Ceftriaxone plus azithromycin (Active Comparator): Single dose ceftriaxone 1 g plus single-dose azithromycin 2 g
  Interventions: Drug: Ceftriaxon; Drug: Azithromycin

INTERVENTIONS:
Drug: Cefixime — Two 400 mg tablets will be administered orally to equal a 800 mg dose.
  Other Names: Cefixime (ATC code J01DD08)
  Arms: Cefixime plus doxycycline
Drug: Doxycyclin — One 100 mg tablet will be administered orally twice a day for 7 days
  Other Names: Doxyhexal (ATC code J01AA02)
  Arms: Cefixime plus doxycycline
Drug: Ceftriaxon — Dose of 1 g intramuscular one time
  Other Names: Ceftriaxone (ATC code J01DD04)
  Arms: Ceftriaxone plus azithromycin
Drug: Azithromycin — Four 500 mg tablets will be administered orally to equal a 2 g dose.
  Other Names: Sumamed (ATC code J01FA10)
  Arms: Ceftriaxone plus azithromycin

SUMMARY:
A non-inferiority, open-label, multicentre randomised controlled trial to compare two therapeutic regimens for the treatment of uncomplicated urogenital, rectal or pharyngeal gonorrhoea in men and women between 18 and 75 years of age. Patients were enrolled and treated from April 2021 to June 2022 at the Dermatovenerology Department, University Hospital Bulovka, Prague, Czech Republic and the Venereology Prague, Medicentrum Beroun, Prague, Czech Republic.

DETAILED DESCRIPTION:
Non-inferiority, open-label, multicentre randomised clinical trial (RCT) compared two regimens for the treatment of uncomplicated urogenital, rectal or pharyngeal gonorrhoea in men and women between 18 and 65 years of age. Patients were enrolled and treated from April 2021 to June 2022 at the Dermatovenerology Department, University Hospital Bulovka, Prague, and the Venereology Prague, Medicentrum Beroun, Prague, Czech Republic.

Laboratory testing The diagnosis of gonorrhoea and C. trachomatis infection was established from urogenital, rectal and pharyngeal swab specimens. Laboratory testing for inclusion in the study and at 3 weeks after initiation of treatment was performed using the Cobas 4800 CT/NG NAAT assay (Roche Diagnostics, Indianapolis, IN, USA). At test of cure visits 1 and 3 weeks after the initiation of treatment, swabs for cultivation of N. gonorrhoeae were also sampled and immediately inoculated onto non-selective and selective Modified Thayer-Martin agar plates. Inoculated agar plates were directly transferred to the hospital laboratory for incubation at 36°C in a humid 5% CO2-enriched atmosphere for 48 hours. Suspected gonococcal colonies were species verified using the biochemical NEISSERIAtest® (LACHEMA, Brno, Czech Republic) or the PolyViteX VCAT3® medium (Biomérieux, Marcy l'Etoile, France).

Statistical analyses Sample size was based on assessing non-inferiority of the cefixime plus doxycycline arm compared to the ceftriaxone plus azithromycin arm with a one-sided 5% type I error rate. We estimated the sample size based on estimates from other gonorrhoea treatment studies and expert opinions. The target sample size of 152 participants (76 per group) was based on an assumed treatment failure of 0% in the ceftriaxone-azithromycin arm and 2% in the cefixime-doxycycline arm, which would provide at least 90% power for the comparison of the primary endpoint. Intention-to-treat (ITT) and per-protocol analyses were done; per protocol results are reported here and ITT results in the online supplement. The ITT population was composed of all randomised patients; the per-protocol population consisted of patients who were randomised, received the allocated regimen (for doxycycline, at least ≥85% (12/14) of the prescribed dose) underwent follow-up examinations, and abstained from any sexual activities, including protected intercourse, during the study period. For each study group, the proportion of patients with urogenital, rectal or pharyngeal gonorrhoea who achieved microbiological cure was calculated. The Clopper-Pearson exact method was used to estimate confidence intervals (CIs). We used chi-square tests (Pearson's or Fisher's test when less than five observations) for binomial outcome measures and Student's t test for continuous outcome measures, as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* uncomplicated urogenital, rectal or pharyngeal gonorrhoea diagnosed using the nucleic acid amplification test

Exclusion Criteria:

* any antimicrobial treatment during the 4 weeks before study enrolment
* pregnancy or lactation
* autoimmune disease
* renal, hepatic or cardiac insufficiency
* immunosuppressive therapy
* allergy to cephalosporins, macrolides or doxycycline

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Number of Participants with negative cultures 1 and 3 weeks and a negative NAAT 3 weeks (±3 days) after treatment initiation. | One and three weeks (±3 days)
  To assess the eradication rate of Neisseria gonorrhoeae by culture and NAAT following a single-dose cefixime 800 mg plus doxycycline 100 mg b.i.d. for 7 days compared to single-dose ceftriaxone 1 g plus single-dose azithromycin 2 g (Intent to Treat population).

SECONDARY OUTCOMES:
Number of Participants with clinical cure defined as disappearance of clinical symptoms and signs 1 week after treatment according to the clinical assessment of the patient by the physician. | One week (±3 days)
  To assess clinical cure (disapperance of clinical symptoms and sings) following a single-dose cefixime 800 mg plus doxycycline 100 mg b.i.d. for 7 days compared to single-dose ceftriaxone 1 g plus single-dose azithromycin 2 g (Intent to Treat population).
Occurrence of treatment-related severe adverse events in treatment groups | One and three weeks (±3 days)
  Adverse event frequency and severity will be compared between patients who received single-dose cefixime 800 mg plus doxycycline 100 mg b.i.d. for 7 days compared to single-dose ceftriaxone 1 g plus single-dose azithromycin 2 g

CONTACTS AND LOCATIONS:
Overall Officials: Filip Rob, MD, PhD, Principal Investigator — Nemocnice Na Bulovce
Locations (2):
- Czechia (2):
  - Venereology Prague, Medicentrum Beroun, Prague
  - University Hospital Bulovka, Prague

IPD SHARING:
Plan to Share IPD: No